CLINICAL TRIAL: NCT02850003
Title: A Phase 1b Open-Label Study Evaluating the Absorption and Systematic Pharmacokinetics of Topically Applied IDP-120 Gel in Subjects With Acne Vulgaris Under Maximal Use Conditions
Brief Title: Absorption and Systematic Pharmacokinetics of Topically Applied IDP-120 Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V01-120A-501
Record Dates: First submitted 2016-07-06; First posted 2016-07-29 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IDP-120 Gel (Experimental): Gel
  Interventions: Drug: IDP-120 Gel

INTERVENTIONS:
Drug: IDP-120 Gel — Gel
  Other Names: Gel

SUMMARY:
Study designed to assess the safety and plasma PK of tretinoin and its metabolites from topically applied IDP-120 gel.

DETAILED DESCRIPTION:
An Open-label study designed to assess the safety and plasma PK of tretinoin and its metabolites from topically applied IDP-120 gel.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between the ages of 9 and <17 (16 years 11 months)
* Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or legal guardian must sign the informed consent.
* Subject must have a score of 3 (moderate) or 4 (severe) on the Evaluator's Global Severity assessment.
* Subject with facial acne inflammatory lesion count no less than 20 but no more than 40.
* Subject with facial acne non-inflammatory lesion count no less than 20 but no more than 100.

Key Exclusion Criteria:

* Use of an investigational drug or device within 30 days of enrollment, previous participation in a research study with IDP-120 Gel, or participation in a research study concurrent with this study.
* Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobate, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram-negative folliculitis.
* Any underlying disease or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion counts inconclusive.
* Subjects with a facial beard or mustache that could interfere with the study assessments
* Subjects with more than 2 facial nodules.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Evaluators Global Severity Score At Day 15 | 15 Days
  Acne severity will be determined by the investigator/evaluator based on the global assessment of the inflammatory and non-inflammatory lesions of facial acne. Evaluations will be graded on a static scale ranging from 0 (clear) to 4 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals
Locations (1):
- Valeant Site 01, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No